CLINICAL TRIAL: NCT04141059
Title: Effect of a French Maritim Pine Bark Extract Oligopin® on Skin Ageing. Double Blind, Parallel, Randomized, Placebo Controled Intervention Trial
Brief Title: Effect of Oligopin® on Skin Ageing
Acronym: OLIGOSKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Fundació Eurecat (Other); Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other); Les Dérivés Résiniques et Terpéniques (DRT) S.A.S. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OLIGOSKIN
Record Dates: First submitted 2019-10-17; First posted 2019-10-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Skin Aging
Keywords: Photoaging; Polyphenols; Natural extracts; Collagen metabolism
MeSH Terms: interventions — Oligopin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oligopin (Experimental): Intervention group that will intake 100 mg of Oligopin® for 6 weeks
  Interventions: Dietary Supplement: Oligopin
- Placebo (Placebo Comparator): Placebo group that will intake 250 mg of Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oligopin — Oligopin capsules composition is :100 mg Oligopin®, 150 mg Maltodextrin, 1.5 mg Mg stearate.
  Arms: Oligopin
Dietary Supplement: Placebo — Placebo capsules composition is: 250 mg Maltodextrin and 1.5 mg Mg stearate
  Arms: Placebo

SUMMARY:
Extrinsic or exogenous ageing is caused by repetitive exposure of the skin to harmful agents, while primary cause the exposure to ultraviolet (UV) radiation, known as photoageing, including solar effect. Chronic solar UV exposure has multiple damaging effects on skin, such as wrinkling, dryness, dyspigmentation, epidermal thinning and increasing fragility. In addition, solar exposure and age increase a subepidermal band.

Fibrillar collagen, which is synthesized from fibroblasts, is the predominant extracellular matrix (ECM) component of the dermis. Collagen type I and III are considered to be the major interstitial, fiber forming collagen in normal human dermis. In addition, the dermis contains collagen types IV (gelatine), V and VI. Other important component of the EMC of the dermis are elastic fibers being elastin (ELN) their main component and play a critical role in skin elasticity and the reduction of elastic fiber production results in impaired elasticity. UV radiation induces ECM degeneration and consequently an increase in fragility and loss of elasticity of the skin. This process is mediated by an increase in matrix metalloproteinases (MMPs) expression in human skin which are responsible for degrading ECM proteins, such as collagen, fibronectin and elastin. The natural inhibitors of MMPs are tissue inhibitors of metalloproteinases (TIMPs), being TIMP-1 the most relevant TIMP affecting collagen metabolism.

DETAILED DESCRIPTION:
Orally administered ingredients can have positive effects on skin characteristics by modulating the internal factors leading to the changes associated with photoageing. Thus, the use of food ingredients and supplements that claim to reduce the risk of skin disorders or alleviate skin ageing is increasing.

Between these ingredients, polyphenols obtained from botanical extracts has been used for cosmetic applications, including Pycnogenol®, a French Maritime Pine Bark extract (FMPBE). showing photoprotective effect against UV-light induced skin damages, and an improvement in hydratation and elasticity of skin in human clinical trials. In another clinical trial, treatment with a different FMPBE called Flavangenol®, significantly decreased skin photo-aged scores. Other human intervention studies with oral administration of polyphenol extracts of different origins such as citrus extract (NutroxSun®), red orange fruit extract (Red Orange Complex®), Polypodium leucotomos and Pomegranate extracts (PPmix® and Fernblock®) have demonstrated beneficials effects of these supplements on improvement of skin characteristics.

The results of the studies cited above suggest that oral administration of polyphenols rich extracts and especially of FMPBE is a promising approach for nutritional photoprotection of skin, reducing photoageing.

Nevertheless, it must be taken into account that most of these studies have been done with a low number of subjects, with combination with other ingredients and/or without placebo group. Thus, well designed clinical trials with a correct volunteer's number are required to obtain robust results about the effects of FMPBE on skin ageing.

Dérivés Résiniques et Terpéniques (DRT) is a company that has developed and commercialize Oligopin®, a polyphenol extract derived from French maritime pine bark. Oligopin® is characterized by a practical absence of tannins ( < 1%) and a high content in low molecular weight oligomeric procyanidins (OPC > 70%; dimers about 20%), a distinctive feature of other proanthocyanidin-rich extracts such as Pycnogenol® which contained about 5% of dimers.

Furthermore, although the insoluble products in water are low in both products, lower and more adequate concentrations are present in Oligopin® (Oligopin ® typically 2 to 4% to a maximum at 5% versus Pycnogenol®: 6% - 8.1%).

The degree of polymerization of OPC can determine its absorption across cell membranes and, as it has been observed in rats, only a certain OPC of a lower degree of polymerization is absorbed during transit in the gut. Consequently, the effect of FMPB extract could be determined, in part, by the quality of its OPC.

The hypothesis of the present study is that circulating metabolic fraction of Oligopin® might exert beneficial actions on collagen metabolism, which is directly linked to skin strength and elasticity.

In consequence, the daily consumption of Oligopin® will exert beneficial effects on skin ageing through the modulation of the proteins involved in the metabolism of collagen in humans.

The main objective of the study is to determine the beneficial effects of Oligopin® on skin aging, through the improvement of skin elasticity in participants with photo-aging.

The secondary objectives of the study are:

* To evaluate the effects of Oligopin® on skin aging through the measurement of wrinkles, spots, skin hydration and subepidermal band.
* To evaluate the effects of Oligopin® on the dynamics of collagen and elastin through the determination of different biomarkers in serum and the expression of genes in peripheral blood mononuclear cells (PBMCs).
* To discover new biomarkers of the effects of Oligopin® through transcriptomic analysis in PBMCs and serum metabolomic analysis.
* To characterize the metabolites of Oligopin® (MFO) in plasma.
* To establish potential correlations between specific metabolites of MFO and the beneficial effects of Oligopin® on the skin, as well as between serum biomarkers and PBMC.
* To evaluate the ability of the MFO to modulate the dynamics of collagen through the use of cellular models of human fibroblasts.

In an initial phase, an acute postprandial study will be carried out with 20 of the 60 volunteers with the consumption of 700 mg of Oligopin® in a single day, with the aim of obtaining the MFO. With MFO, the mechanisms by which Oligopin® exerts the beneficial effects on skin aging will be studied through in vitro studies with cellular models. The 60 participants will participate in the second phase of the study, which will be randomly divided into two groups of 30 participants, depending on whether they consume a 100 mg Oligopin® capsule or a placebo capsule, with the same appearance as the Oligopin® capsule but will not contain the botanical extract. In this second phase, participants will consume one capsule each day for a total of 6 weeks.

During the study there will be 5 visits, one of selection (V0), one of the first phase of the study (V1; week 1) and 3 visits of the second phase of the study (V2, V3 and V4; weeks 2, 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

* Men and women 35 years or more age.
* Fitzpatrick skin phototype II-IV.
* Signed informed consent.

Exclusion Criteria:

* Present intolerances and/or food allergies related to Oligopin®.
* Being pregnant or intending to become pregnant.
* Be in breastfeeding period.
* Be a smoker.
* Participate in or have participate in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
* Present some chronic gastrointestinal disease.
* Present some chronic disease with clinical manifestation.
* Receive or are planning to receive facial cosmetic procedures such as facial peel, dermabrasion, laser treatments within six months prior to start the study.
* Take supplements or multivitamin supplements or phytotherapeutic products that interfere with the treatment under study up to 30 days before the start of the study.
* Has or are planning to take acne treatments, photoaging treatments or topical prescription products indicated for improving the appearance or condition of skin within 30 days.
* Present any skin disease (e.g., atopic skin, eczema, neurodermatitis or psoriasis) or other dermatological disorders (e.g., scars, sunburn or moles).
* Intensive sun or artificial UV exposure (solarium) on the test area within 30 days prior to study start or planned during the study period.
* Being unable to follow the study guidelines.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Change in skin elasticity | At weeks 2, 3 and 4
  Skin elasticity measured by using a Cutometer® MPA 580

SECONDARY OUTCOMES:
Change in skin wrinkles | At weeks 2, 3 and 4
  Skin wrinkles measured using DermoPrime System
Change in skin hydratation | At weeks 2, 3 and 4
  Skin hydratation measured using DermoPrime System
Change in skin spots | At weeks 2, 3 and 4
  Skin spots measured using DermoPrime System
Change in subepidermal low-echogenic band | At weeks 2, 3 and 4
  Subepidermal low-echogenic band measured by ultrasound echogenicity quantitative approach
Change in biomarkers of collagen and elastin dynamics in serum | At weeks 2 and 4
  Serum levels of Human Procollagen I N-Terminal Propeptide, Human Procollagen I C-Terminal Propeptide, Human C-Telopeptide of Type I Collagen, Fibronectin, Elastin, Hyaluronic acid, MMP-1, TIMP-1. These biomarkers will be measured using humans ELISA kits.
Change in expression levels of genes related to collagen synthesis and degradation in PBMCs | At weeks 2 and 4
  Expression levels in PBMCs by quantitative polymerase chain reaction (qPCR) of the following genes: Collagen type I alpha 1 chain gene (Col1a1), Collagen type I alpha 2 chain gene (Col1a2), Mmp-2, Timp-1.
Oligopin® long-term blood metabolites characterization | At weeks 2 and 4
  Oligopin® blood metabolites will be measured by liquid chromatography quadruple Time-of-Flight (LC-qTOF). It will be analyzed the correlations between specific Oligopin® metabolites and its effects on skin, as well as on serum and PBMCs biomarkers.
Transcriptomics in PBMCs | At weeks 2 and 4
  Transcriptomics in PBMCs analyzed using microarrays Agilent technologies
Metabolomics in serum | At weeks 2 and 4
  Non-targeted metabolomics of aqueous and lipid fraction of serum samples measured using proton nuclear magnetic resonance
Postprandial Oligopin® blood metabolites characterization | At week 1
  Postprandial Oligopin® blood metabolites characterization after 700 mg Oligopin® consumption and measured by LC-qTOF. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to modulate collagen levels | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of total collagen concentration in cells and cultured media. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to modulate secreted collagen type I | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of secreted collagen type I. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to modulate secreted collagen type III | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of secreted collagen type III. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to modulate pyruvate target genes | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of mRNA levels of pyruvate target genes in cells measuring expression levels of elastin, Col1a1, Col1a2, Col3a1, Mmp-1 and Timp-1 genes. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to modulate MMP-1 activity | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of MMP-1 activity in culture medium. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to modulate TIMP-1 levels | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of TIMP-1 levels in culture medium. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to inhibit MMP-1 activity | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of inhibitory effect on MMP-1. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to inhibit MMP-2 activity | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of inhibitory effect on MMP-2. The measurements will be done at 0 hours, 2 hours and 6 hours.
Capacity of Oligopin® blood metabolites to inhibit MMP-9 activity | At week 1
  The capacity of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of inhibitory effect on MMP-9. The measurements will be done at 0 hours, 2 hours and 6 hours.
Effect of Oligopin® blood metabolites on collagen fibers cross-linking | At week 1
  The effect of Oligopin® blood metabolites to modulate collagen dynamics using human fibroblast cell line treated with Oligopin® blood metabolites and determination of collagen fibers cross-linking effect. The measurements will be done at 0 hours, 2 hours and 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Dr, Principal Investigator — UTNS (Eurecat_Reus)/HUSJR. Reus, Tarragona, Spain.
Locations (1):
- Centro Tecnológico de Nutrición y Salud (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org